CLINICAL TRIAL: NCT01193374
Title: Promoting Healthy Families Through Enhanced Primary Care
Brief Title: The Healthy Families Project
Acronym: HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Ardis L. Olson, Dartmouth College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21HD050996 (NIH)
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Childhood Obesity
Keywords: Childhood Obesity; Primary Care; Counseling; Screening
MeSH Terms: conditions — Pediatric Obesity | interventions — Counseling; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent/child tailored mailed materials (Experimental): Family provided newsletters tailored to issues and readiness to change. Family receives educational nutrition DVD, pedometers for family activities and child nutrition/physical activity games
  Interventions: Behavioral: Clinician enhanced screening and counseling prompts; Behavioral: Tailored education and motivational materials
- Basic information at single time (Active Comparator): Family provided with high quality booklet from American Dietetic Association providing the same information that intervention arm received but not tailored.
  Interventions: Behavioral: Clinician enhanced screening and counseling prompts; Behavioral: basic educational brochure

INTERVENTIONS:
Behavioral: Clinician enhanced screening and counseling prompts — PDA based health risk screening for well child issues and obesity risks
  Other Names: All subjects receive screening/counseling
Behavioral: Tailored education and motivational materials — Specific tailoring for those interested in change vs not . Two newsletters over 3 mpn.
  Other Names: Well child care intervention
  Arms: Parent/child tailored mailed materials
Behavioral: basic educational brochure — Booklet by ADA sent x 1.
  Other Names: Education
  Arms: Basic information at single time

SUMMARY:
A primary care approach to obesity prevention will be developed and tested in a randomized trial in 4 pediatric primary care practices. Enhanced screening for obesity risks and prompts for effective counseling at well visits of 4 to 10 year olds will be developed utilizing hand held technology( PDAs). The impact on the content and quality of clinician counseling will be assessed in exit survey prior to and after implementation. Among families interested in making a change to address nutrition or activity risk reported on the screener a cohort with children > BMI 85% will be recruited. They will be randomized to mailed tailored supports to level of readiness to change versus a single generic informational mailing. The hypotheses are that 1)families that receive the enhanced office visit with screening will be more likely to plan to make changes compared to usual care; and 2) families receiving the tailored post visit supports will be less likely to gain weight than controls after 6 months.

DETAILED DESCRIPTION:
1. Using hand held PDAs, we will develop an obesity risk screening and counseling system for 4 through 10 year olds attending primary care well child visits. Screening results will be summarized immediately by the PDA and will prompt the clinician to provide brief counseling messages tailored to each childís obesity screening results, including the familyís and the childís readiness to change behavior
2. We will evaluate the specific content and quality of clinician obesity counseling provided at the well child visit through parent surveys before and after implementation of the PDA screening and counseling program.
3. To support action by families after the office visit, we will develop a post-visit intervention package of newsletters and materials that are tailored to child/family obesity risk behaviors and parental readiness to change.
4. We will evaluate the impact of this post visit intervention program in a 6 month trial focused on children identified at well child screening to have BMI >85%. 200 Families will be randomized to receive either a series of mailed supports over 3 months versus a single generic-content mailing. We will determine the respective impact of these two levels of post-visit support on stage of change, parental action on key obesity risk behaviors, and stabilization of BMI z scores after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Families with children ages 4 to 11 years
* For post visit supports; Children > 85% for age BMI

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2007-02; Primary Completion 2008-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
BMI z score | 6 months
  Prevention of increase in BMI

SECONDARY OUTCOMES:
Parental readiness to initiate change | immediately post well visit
  Exit surveys comparing parents with PDA screening vs not for readiness to make changes

CONTACTS AND LOCATIONS:
Overall Officials: Ardis L Olson, MD, Principal Investigator — Dartmouth Medical School, Dept. of Pediatrics
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Dartmouth Medical School, Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire